CLINICAL TRIAL: NCT04493489
Title: Propranolol Adjuvant Treatment of Bladder Cancer: a Randomized Phase II Clinical Trial
Brief Title: Propranolol Adjuvant Treatment of Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Yijing He, Associate Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020/prop/bladder/CSU
Record Dates: First submitted 2020-07-24; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCG (Placebo Comparator): After TURBT, the first year: once a week for 6 times, from the 7th week, once every 2 weeks, and 3 times. Administer once a month starting from the 13th week and continue to give 10 times. Second and third years: once a month, 12 times a year.
  Interventions: Drug: BCG
- Propranolol plus BCG (Experimental): After TURBT administered for 2 consecutive years, oral propranolol, starting dose 10mg, tid, then 20mg, tid,lastly increased to 40mg, bid. After the last BCG infusion, propranolol was gradually reduced, in the order of 20 mg, tid to 10 mg, tid.
  Interventions: Drug: Propranolol Hydrochloride; Drug: BCG

INTERVENTIONS:
Drug: Propranolol Hydrochloride — Trial group: BCG + propranolol: after TURBT administered for 2 consecutive years, oral propranolol, starting dose 10mg, tid, then 20mg, tid,lastly increased to 40mg, bid. After the last BCG infusion, propranolol was gradually reduced, in the order of 20 mg, tid to 10 mg, tid.
  Arms: Propranolol plus BCG
Drug: BCG — Control group: BCG vaccine: After TURBT, the first year: once a week for 6 times, from the 7th week, once every 2 weeks, and 3 times. Administer once a month starting from the 13th week and continue to give 10 times. Second and third years: once a month, 12 times a year.

SUMMARY:
Bladder cancer (bladder cancer) is the tenth most common cancer in the world, ranking 13th in the number of deaths. There are about 549000 new cases of bladder cancer worldwide, with 200000 deaths and a higher incidence rate in men than in women. In 2013, the incidence rate of bladder cancer was high in China, accounting for 2.02% of all new cases. Bladder cancer has become a major disease threatening people's life and health. Therefore, the exploration of the mechanism of the occurrence and development of bladder cancer and effective drugs has been an important focus of bladder cancer research. The current treatment of bladder cancer is mainly TURBT (transurethral resection of bladder tumour) resection and BCG, chemotherapy adjuvant treatment, but its recurrence and metastasis still exist, so this study aims to explore an effective drug treatment. The purpose of this study was to investigate the safety and efficacy of propranolol in adjuvant BCG therapy, and whether propranolol can effectively alleviate the metastasis and recurrence of bladder cancer and improve the survival time after bladder cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 75
2. Patients with pathologically confirmed non-muscle invasive bladder cancer (T1 / Ta high grade / CIS), according to the 2004 WHO classification criteria
3. No evidence of patients with muscular invasive disease
4. American Oncology Group ECOG score <2
5. Patients' expected survival time should be more than 3 months
6. Organ function and hematopoietic function must meet the following requirements: hemoglobin (HGB) ≥ 90g / L; white blood cell count (WBC) ≥ 3 × 10 ^ 9 / L; absolute neutrophil count (ANC) ≥ 1.5 × 10 ^ 9 / L Platelet count (PLT) ≥100 × 10 ^ 9 / L; total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase ( ALT) ≤ 2.5 × ULN; if abnormal liver function is due to tumor liver metastasis, AST or ALT ≤ 5 × ULN; serum creatinine (Cr) ≤ 1.5 × ULN; international standardized ratio (INR) or plasma prothrombin time PT) ≤1.5 × ULN
7. Blood pressure with acceptable surgery: blood pressure greater than 90 / 60mmHg, resting heart rate greater than 60 beats / min
8. Volunteer to participate in clinical research; fully understand, inform, and sign the consent form; willing to follow and have the ability to complete all test procedures

Exclusion Criteria:

1. Contraindications for propranolol: bronchial asthma, cardiogenic shock, cardiac block (II-III degree Atrioventricular conduction block), severe or acute heart failure, sinus bradycardia
2. In use or have used any beta-blockers for disease reasons in the past two years
3. Patients with other malignancies within 5 years before enrollment, in addition to cervical carcinoma in situ and cured skin basal cell carcinoma with appropriate treatment
4. Immunodeficiency, such as patients with HIV infection or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation
5. Patients with tumor brain metastases and bone marrow metastases were excluded, and patients with liver metastases and lung metastases could be included
6. Participants who have participated in clinical studies of drugs other than BCG within 4 weeks
7. Patients with a history of allergy to propranolol
8. Alcohol, drug or substance abuse history in the past year
9. Subject has an active infection or an unexplained fever during screening, before the first dose> 38.5 degrees(According to the researcher's judgment, the subjects can be enrolled due to the fever caused by the tumor)
10. Any situation that the investigator believes may increase the risk of the subject or interfere with clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2020-09-06 (Estimated); Primary Completion 2023-09-06 (Estimated); Study Completion 2024-09-06 (Estimated)

PRIMARY OUTCOMES:
two-year recurrence-free survival | 24 months